CLINICAL TRIAL: NCT05427929
Title: A Pilot Study of Measuring Diaphragm Electrical Activity in Neonates Using a Smaller Inter-electrode Distance
Brief Title: Measuring Diaphragm Electrical Activity in Neonates Using a Smaller Inter-electrode Distance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 21-0224-A
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Distress Syndrome, Newborn; Infant, Premature
Keywords: Preterm Neonates; NAVA Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NVR 4mm Edi Catheter (Experimental)
  Interventions: Device: NVR 4mm Edi catheter

INTERVENTIONS:
Device: NVR 4mm Edi catheter — Receive NAVA ventilation using the newly designed NVR 4 mm Edi catheter

SUMMARY:
Neurally Adjusted Ventilatory Assist (NAVA) is a mode of ventilation where the electrical activity of the diaphragm (EDI) - a signal representing the baby's respiratory drive - is used to control the timing and amount of assist provided. NAVA was introduced to the market in 2007 and since has been used in more than 40 countries.

In the current clinical practice, the Edi signal from the patient is captured with miniature sensors (the size of a hair) embedded in the wall of a specially designed naso/orogastric feeding tube. This FDA and Health Canada approved, commercially available catheter (Getinge, Solna, Sweden), is 6 Fr in size (outer diameter), 49 cm in length and has 8 pairs of sensors that are placed 6 mm apart (so-called inter electrode distance (IED) is 6 mm).

While no obvious side effects have been noted by clinicians, for the smallest of neonates, the currently used commercial catheter (size 6F, 49 cm long) may have 'excessive' post-array catheter length. In these neonates, typically those with weight < 1000 grams, following the correct placement of catheter as per the electrode array positioning at gastro-esophageal junction, the feeding holes in the catheter may end at the level of distal stomach instead of the desirable mid-stomach location. The changing demographics of the patients in the Neonatal Intensive Care Units (NICU) has created a clinical need to redesign the currently used Edi catheter specifically to suit the smallest of patients, such that following adequate placement the feeding holes sit at the level of mid-stomach. Drs. Christer Sinderby and Jennifer Beck in Toronto, Canada, are the original designers of the 6 mm/49 cm currently used Edi catheter. These investigators (at St-Michael's Hospital, Toronto) in collaboration with their team at Neurovent Research Inc. (NVR) have re-designed and invented a new prototype of the current FDA-approved catheter specifically suited for use in extreme premature neonates. They have done so by reducing the interelectrode distance from the originally set 6 mm to 4 mm, which reduces the overall insertion depth to capture the same signal from the diaphragm. All other parameters are exactly same as the original catheter (6F, 49 cm long).

In this small feasibility study the investigators wish to provide a clinical proof of concept for the use of this newly designed prototype in 10 extremely premature neonates who are already receiving NAVA ventilation in the NICU.

DETAILED DESCRIPTION:
This is an unblinded pilot study to evaluate the performance of the new 4 mm IED. The procedures required for this evaluation include placement of the new NVR 4 mm Edi catheter, and ventilation in the NAVA mode. All these procedures are considered to have no significant additional risk. Supervision by a physician or respiratory therapist with expertise in Edi catheter and NAVA will be present, in line with the current clinical practice in the Mount Sinai NICU.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with current weight <1000g who are already receiving invasive or non-invasive NAVA ventilatory support using the standard 6 mm IED Edi catheter will be eligible for recruitment.

Exclusion Criteria:

* Infants deemed to be unstable by the attending clinician from a respiratory or hemodynamic perspective
* Known congenital or chromosomal anomalies
* Any acute illness such as sepsis, necrotizing enterocolitis or acute pulmonary hypertension
* Parental consent not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of re-initiating NAVA ventilation with new NVR 4mm Edi Catheter | During study catheter change (total study length = 2 hours during procedure)
  Categorical (yes/no) - Feasibility will be defined as 4mm catheters picking up EDI signals and allowing initiation of NAVA ventilation as per the standard clinical practice. Cases where clinical team is unable to initiate NAVA, necessitating change back to 6 mm catheters will be termed non-feasible.

CONTACTS AND LOCATIONS:
Overall Officials: Amish Jain, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada